CLINICAL TRIAL: NCT05258175
Title: Effects of Thoracic Kinesiotaping on Pulmonary Function and Functional Capacity of COPD Patients
Brief Title: Effects of Kinesiotaping Technique on Lung Function & Functional Capacity of Chronic Obstructive Lung Disease Patients
Acronym: COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Umra Ihsan
Record Dates: First submitted 2022-02-20; First posted 2022-02-28 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; Functional capacity; Pulmonary function; Thoracic Kinesiotaping
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Masking Description: single
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio taping muscle facilitation technique along with standardized physiotherapy protocol (Experimental): On the diaphragmatic muscle, muscle facilitation technique will be applied from proximal to distal with 10-15% tension when the participant is standing and exhaled out and the body is in extension. The base of the tape will be about 1 inch below the xiphoid area.
  Then the one tail of tape applied with 10% tension on the rib cage with maximum deep inspiration followed by expiration and the other tail of tape will be applied to the subcostal area in forward bending position while taking deep breath with arms adduct and being crossed.
  The tape will be changed on every fifth day and assessment will be done at baseline and 2nd week of intervention Total number of sessions: 3
  Interventions: Other: KT; Other: Standardized physiotherapy protocol
- Standardized physiotherapy protocol (Active Comparator): Pursed lip breathing exercise: Patient instructed to breathe through nose and inspiration should be slowly and expiration is done through mouth by pursing the lips slowly such that if flame is held in front, then the flame should be bended but not blow off. 3 sets a day for 15 days.
  Diaphragmatic breathing exercise: Patient sitting comfortably, with knees bent and shoulders, head and neck relaxed. Patient will be instructed to place one hand on upper chest and the other just below your rib cage. Breathe in slowly through nose so that stomach moves out against your hand. 3 sets a day for 15 days.
  Deep breathing exercise: Patient instructed to take "slow and deep breaths, inhaling through the nose and exhaling through the mouth". Participant is asked to place their hand on their abdomen and expand their abdomen to lift their hand during inhalation. 3 sets a day for 15 days.
  Interventions: Other: Standardized physiotherapy protocol

INTERVENTIONS:
Other: KT — Kinesio tapping will be applied in three session and it will be changed on every fifth day in total 15 days.
  Arms: Kinesio taping muscle facilitation technique along with standardized physiotherapy protocol
Other: Standardized physiotherapy protocol — 3 sets with five repetitions per day for total of 15 days.

SUMMARY:
This study is designed to determine the effects of diaphragmatic kinesiotaping (KT) facilitation technique on pulmonary function, functional capacity and forward head posture of chronic obstructive lung diseases (COPD) patients. The application of KT as an adjunct to conventional protocol in COPD patients if proven effective can enhance the symptom control in COPD patients for improving lung function, posture reducing the perception of dyspnea as well as improving functional capacity.

DETAILED DESCRIPTION:
The Global Initiative for Chronic Obstructive Lung Disease 2019 report defines Chronic Obstructive Pulmonary Disorders (COPD) as a "common, preventable and treatable disease that is characterized by persistent respiratory symptoms and airflow limitation that is due to airway or alveolar abnormalities, usually caused by significant exposure to noxious particles or gases". COPD is one of the leading causes of morbidity and mortality and will become the third leading cause of death and the fifth commonest cause of disability in the world. The airway obstruction in COPD cause mechanical disadvantage and increased respiratory work and dyspnea symptoms, limitations in exercise, and reduced Physical Activity Level. Patients with COPD experience muscle wasting particularly of skeletal muscle and also shortens the length of inspiratory muscles, particularly the diaphragm, resulting in functional muscle dysfunction and weakness which then results in a reduction in functional capacity, quality of life.

Different managements for COPD are provided in the literature, which includes bed rest, pharmacological therapy, oxygen therapy, and physical therapy. Physical therapy management include breathing exercises and early mobilization to restore or maintain muscle function in COPD stages. Kinesiotaping is relatively new band aid method used worldwide for the treatment of musculoskeletal disorder symptoms. Kinesiotaping applied on certain region stimulate proprioceptive awareness and re educate the patient to adopt its normal posture during their normal life activity and thus normalize the muscles overactivity in the patients. KT is said to promote the respiratory muscle activation specifically the diaphragm muscle and also reduce the tension on muscle.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed patients of COPD falling in stage I-III according to The Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria.
* GOLD 1 -mild: Forced Expiratory Volume in 1 sec (FEV1) ≥80%, GOLD 2 - moderate: 50% ≤ FEV1 <80% predicted and GOLD 3 - severe: 30% ≤ FEV1 <50% predicted
* Age between 40-70 years.
* Both genders
* Volunteering to participate in study

Exclusion Criteria:

* COPD exacerbation within last 4 weeks
* Allergic reaction to the taping material,
* Patients with recent chest wall trauma, surgery, deformity having scar, lesion, or incision in area of KT application.
* Uncontrolled arterial hypertension and diabetes mellitus.
* Patients with neurological, musculoskeletal, cardiac, pulmonary disease with physical impairment and history of psychiatric illness

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
Peak expiratory flow rate (PEFR) Peak expiratory flow rate (PEFR) | 15 days
  Peak expiratory flow rate (PEFR) Peak expiratory flow rate (PEFR) measured through digital spirometer. Peak Expiratory Flow Rate (PEFR) measured through digital spirometer. Three zones of measurement are commonly used to interpret peak flow rates. Normal value of PEFR is (80-100%). Green zone indicates 80 to 100 percent of the usual or normal peak flow reading, yellow zone indicates 50 to 79 percent of the usual or normal peak flow readings, and red zone indicates less than 50 percent of the usual or normal peak flow readings.
  Changes in PEFR from baseline to 5th and after 15th day of intervention will be assessed.
Forced vital capacity (FVC) | 15 days
  Forced vital capacity (FVC) measured through digital spirometer. If the value of FVC is within 80% of the reference value, the results are considered normal.
  Changes in FVC from baseline to 5th and after 15th day of intervention will be assessed.
Forced expiratory volume in 1sec (FEV1) | 15 days
  Forced expiratory volume in 1sec (FEV1) measured through digital spirometer. If the value of FEV1 is within 80% of the reference value, the results are considered normal.
  Changes in FEV1 from baseline to 5th and after 15th day of intervention will be assessed.
FVC/FEV1 | 15 days
  FVC/FEV1 measured through digital spirometer. The normal value for the FEV1/FVC ratio is 70% (and 65% in persons older than age 65).
  Changes in FVC/FEV1 from baseline to 5th and after 15th day of intervention will be assessed.
Six-minute walk test (6MWT) | 15 days
  The six-minute walk test (6MWT) is a submaximal exercise test for assessing physical functional capacity in patients with COPD.
  It is a test that measures how far a person can walk in 6 minutes. Changes in 6MWT from baseline to 5th and after 15th day of intervention will be assessed.
Modified Medical Research Council Dyspnea Scale (mMRC) | 15 days
  The mMRC dyspnea score is a 5-point (0-4) scale based on the severity of dyspnea.
  0, no breathlessness except on strenuous exercise and and 4, too breathless to leave the house, or breathless when dressing or undressing.
  Changes in mMRC scale from baseline to 5th and after 15th day of intervention will be assessed.

SECONDARY OUTCOMES:
Craniovertebral angle (CVA) | 15 days
  CVA is measured by taking 2 lateral photographs of the subject in a relaxed seated position without a back support. Spinous process of C7 and the tragus of ear are marked with a body marker. A horizontal line is drawn passing through C7 making a right angle with the vertical. Then, the angle between the line connecting C7 spinous process with the tragus of the ear and the horizontal line, is measured using goniometer.
  Craniovertebral angle of less than 50 degrees while standing is commonly considered forward head posture.
  It will be assessed from baseline to 5th day and after 15th day of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Suman Sheraz, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Pak Medical Center Hospital, Peshawar, Khyber Pukhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No